CLINICAL TRIAL: NCT04731454
Title: Feasibility and Acceptability of a Healthy Nordic Diet Intervention for the Treatment of Depression: a Randomized Controlled Pilot Trial
Brief Title: Feasibility and Acceptability of a Healthy Nordic Diet Intervention in Depressed and Non-depressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2020-03735
Record Dates: First submitted 2021-01-16; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Diet; Nutrition; Randomized controlled trial; Pilot study; Healthy Nordic diet
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Nordic Diet (ND) (Experimental): A healthy diet meeting and exceeding the Nordic Nutrition Recommendations and with more than 80% foods from the Nordic region.
  Interventions: Other: Healthy Nordic Diet (ND)
- Control Diet (CD) (Experimental): A control diet approximating the average depressed person's diet, i.e. of somewhat lower quality than the average Swedish diet.
  Interventions: Other: Control Diet (CD)

INTERVENTIONS:
Other: Control Diet (CD) — All food was provided to participants for the duration of the intervention (8 days), including prepared lunches and dinners and ingredients for breakfasts and snacks. A sugar-sweetened juice drink was provided for consumption of one portion per day. Water, milk, coffee, tea and alcohol were consumed as usual.
  Arms: Control Diet (CD)
Other: Healthy Nordic Diet (ND) — All food was provided to participants for the duration of the intervention (8 days), including prepared lunches and dinners and ingredients for breakfasts and snacks. Water, milk, coffee, tea and alcohol were consumed as usual.
  Arms: Healthy Nordic Diet (ND)

SUMMARY:
In the future, we plan to conduct an 8-week diet intervention to investigate whether a healthy Nordic diet improves depression symptoms. The present pilot study tested whether the planned meals and diets were well-liked and accepted by participants (both depressed and non-depressed) in order to ensure that the future diet intervention will be feasible and successful. We also investigated whether any changes in health occurred after 8 days of this diet intervention.

DETAILED DESCRIPTION:
After providing their written informed consent, participants were randomized to receive either a healthy Nordic diet or a control diet for 8 days. All meals were provided and minimal food preparation was required. Participants picked up their food outside the study kitchen every 3 days. Before and after the intervention, health-related self-rated questionnaires were completed. For every meal during the intervention, participants completed a questionnaire on their perceptions of the meal. Every evening a questionnaire was completed to assess dietary adherence. At the end of the study, a final evaluation questionnaire was completed to assess participants' perceptions of the diet and study as a whole.

ELIGIBILITY:
Inclusion Criteria:

* If depressed, a score between 13 and 34 on the Montgomery-Åsberg Depression Rating Scale, self-rated (MADRS-S), indicating mild or moderate depression

Exclusion Criteria:

* A score of 8 or higher (out of a maximum of 12 points) on a brief diet survey (the retired version of the Swedish Food Agency's online Matvanekollen, conducted via phone interview), indicating a relatively healthy habitual diet
* Presence of food allergies, intolerances or sensitivities
* Consuming any form of special diet that excludes certain foods, for example a vegetarian or gluten-free diet
* Suicidality, indicated by a score of 4 or higher on the MADRS-S suicidality question.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Median rating of the liking of all meals as assessed by a Likert item (the Hedonic scale) | 8 days
  1=Dislike very much, and 7=Like very much. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of the appearance of all meals as assessed by an original Likert item | 8 days
  1=Dislike very much, and 7=Like very much. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of the smell of all meals as assessed by an original Likert item | 8 days
  1=Dislike very much, and 7=Like very much. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of the extent to which the smell matches the appearance of the meals as assessed by an original Likert item | 8 days
  1=Doesn't match at all, and 5=Matches very well. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of the taste intensity of all meals as assessed by a Just About Right (JAR) scale | 8 days
  1=Much too low, 3=Just right, and 5=Much too high. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of the portion size of all meals as assessed by a Just About Right (JAR) scale | 8 days
  1=Much too small, 4=Just right, and 7=Much too big. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median rating of feelings of fullness after the meals as assessed by an original visual analog scale (VAS) | 8 days
  0=Not at all full, and 100=Have never felt so full. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Median perception of healthiness of all meals as assessed by an original visual analog scale (VAS) | 8 days
  0=Not at all healthy, and 100=Very healthy. Median of responses for all meals for each participant calculated first, and then the median of those medians calculated and reported for each diet group.
Total amount of non-study foods consumed as assessed by self-report on a questionnaire every evening | 8 days
Total amount of non-study drinks consumed as assessed by self-report on a questionnaire every evening | 8 days
Total amount of provided juice drink not consumed as assessed by self-report on a questionnaire every evening. | 8 days
  Applies to the CD group only.
Rating of how easy it was to follow the protocol, as assessed by an original Likert item on the final questionnaire | 8 days
  1=It was very hard, and 7=It was very easy
Rating of how easy it would be to participate in such a study, with meals recurring every 8 days for 8 weeks (but not having to fill out a questionnaire for the meals) | 8 days
  Assessed by an original Likert item on the final questionnaire where 1=It would be very hard, and 7=It would be very easy

SECONDARY OUTCOMES:
Change in work impairment after 8 days, as calculated from questions of the Work Productivity and Activity Impairment (WPAI) questionnaire | 8 days
  Expressed as percentage impairment, from 0-100%, where higher values indicate greater impairment in work ability
Change in activity impairment after 8 days, as calculated from questions of the Work Productivity and Activity Impairment (WPAI) questionnaire | 8 days
  Expressed as percentage impairment, from 0-100%, where higher values indicate greater impairment in ability to perform daily activities.
Change in gastrointestinal symptom severity after 8 days, as assessed by the total mean score of the Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire | 8 days
  1=no symptoms, 7=very severe symptoms
Change in indigestion symptom severity after 8 days, as assessed by the indigestion sub-score of the Gastrointestinal Symptoms Rating Scale (GSRS) questionnaire | 8 days
  1=no symptoms, 7=very severe symptoms
Change in physical activity level after 8 days, as assessed by the Frändin-Grimby Physical Activity Scale | 8 days
  Score of 1-6, from least to most active
Change in depression severity after 8 days, as assessed by the total score of the Montgomery-Åsberg Depression Rating Scale, self-rated (MADRS-S) questionnaire | 8 days
  Score of 0-54, from least to most severe symptoms
Change in perceived general health status after 8 days, as assessed by the visual analog scale (VAS) question of the EuroQol Health-Related Quality of Life (EQ-5D-5L) questionnaire | 8 days
  0=Worst health imaginable, 100=Best health imaginable
Change in general health after 8 days, as assessed by the summary index value calculated from the questions of the EuroQol Health-Related Quality of Life (EQ-5D-5L) questionnaire | 8 days
  0=health as bad as dead, 1=full health
Self-reported change in health after 8 days, as assessed by a written open-ended response on the final questionnaire | 8 days
  Due to the open-ended, self-reported nature of the responses, they are summarized narratively rather than quantitatively.
Change in body weight after 8 days, as assessed by self-measurement or approximation | 8 days
  Change between self-reported baseline and follow-up body weights calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Sabet, PhD, Study Director — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Närke, Sweden

IPD SHARING:
Plan to Share IPD: No